CLINICAL TRIAL: NCT01112878
Title: Randomized, Double-Blinded, Placebo-controlled Study to Evaluate the Analgesic Efficacy of Oral Clonidine and Gabapentin as Part of a Multi-modal Analgesic Regimen for Preventing Pain After Arthroscopic Shoulder or Knee Surgery
Brief Title: Oral Clonidine & Gabapentin: Improving Recovery and Pain Management After Outpatient With Major Orthopedic Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Several studies going on at the same time.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ronald Wender, Chairman, Department of Anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00019373
Record Dates: First submitted 2010-04-23; First posted 2010-04-29 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Shoulder Arthroscopy; Knee Arthroscopy
Keywords: Shoulder arthroscopy; Knee arthroscopy; Clonidine; Gabapentin; Pain management; Ambulatory surgery; Perioperative outcome; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Sugars; Gabapentin; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugar Pill (Placebo Comparator): Frequency and Dosage:
  * once in the preoperative holding area and once before discharge from PACU
  * continuation of 1 capsule twice daily with meals, 1 to 4 days after surgery.
  Interventions: Drug: Gabapentin; Drug: Clonidine
- Clonidine (Active Comparator): Dosage: 0.2 mg
  * once in the preoperative holding area and once before discharge from PACU
  * continuation of 1 capsule twice daily with meals, 1 to 4 days after surgery.
  Interventions: Drug: Sugar pill; Drug: Gabapentin
- Gabapentin (Active Comparator): Dosage: 600 mg
  * once in the preoperative holding area and once before discharge from PACU
  * continuation of 1 capsule twice daily with meals, 1 to 4 days after surgery.
  Interventions: Drug: Sugar pill; Drug: Clonidine

INTERVENTIONS:
Drug: Sugar pill — Dosage form: capsule, by mouth
  Dosage: not applicable
  Frequency and Dosage:
  * once in the preoperative holding area and once before discharge from PACU
  * continuation of 1 capsule twice daily with meals, 1 to 4 days after surgery.
  Other Names: placebo
  Arms: Clonidine; Gabapentin
Drug: Gabapentin — Dosage form: capsule, by mouth
  Dosage: 600 mg
  Frequency and duration:
  * once in the preoperative holding area and once before discharge from PACU
  * continuation of 1 capsule twice daily with meals, 1 to 4 days after surgery.
  Other Names: Neurontin
  Arms: Clonidine; Sugar Pill
Drug: Clonidine — Dosage form: capsule, by mouth
  Dosage: 0.2 mg
  Frequency and duration:
  * once in the preoperative holding area and once before discharge from PACU
  * continuation of 1 capsule twice daily with meals, 1 to 4 days after surgery.
  Other Names: Catapres
  Arms: Gabapentin; Sugar Pill

SUMMARY:
The purpose of this research is to investigate the non-opioid (non-narcotic) pain-relieving medications clonidine and gabapentin to see if they decrease the amount of opioid pain medications needed after surgery, thereby reducing opioid-related side effects, and time required to return to normal activities of daily living after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo arthroscopic joint surgery
* Willingness and ability to sign an informed consent document
* No allergies to clonidine, gabapentin, anesthetic or analgesic medications
* 18 - 80 years of age
* American Society of Anesthesiologists (ASA) Class I - III adults of either sex
* Women of childbearing potential must be currently practicing an acceptable form of birth control, and have a negative urine pregnancy test

Exclusion Criteria:

* Patients with known allergy, hypersensitivity or contraindications to clonidine, gabapentin, anesthetic or analgesic medications
* Patients with clinically-significant medical conditions, such as brain, heart, kidney, endocrine, or liver diseases, peptic ulcer disease or bleeding disorders
* Patients with chronic hypertension or pain syndromes receiving clonidine or gabapentin, respectively.
* Pregnant or lactating women
* Subjects with a history of alcohol or drug abuse within the past 3 months
* Patients taking any analgesic medications within 48 hours prior to the surgery
* Any other conditions or use of any medication which may interfere with the conduct of the study
* Non-English speakers
* Patients greater than 80 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain using a Verbal Rating Scale (VRS) | 1 month
  Outcomes will be measured with follow up questionnaires at 1, 2, or 3, then 7 and 30 days after surgery

SECONDARY OUTCOMES:
Opioid consumption obtained from the recorded data | 1 month
  Perioperative use of opioid consumption inside hospital (recorded by study staff and data obtained from patient charts) Post discharge use of opioid consumption (data obtained from the follow up questionnaires at 1, 2, or 3, then 7 and 30 days after surgery)
postoperative nausea and vomiting using a Verbal Rating Scale | 1 month
  Outcomes will be measured with follow up questionnaires at 1, 2, or 3, then 7 and 30 days after surgery
return to normal activities of daily living using follow up questionnaires | 1 month
  return to normal activities of daily living(including dietary intake, bowel and bladder function, physical activities)
Patient satisfaction using a verbal rating scale from 0 to 100 | 1 month
  0= Not satisfied 100= Excellent

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Wender, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States